CLINICAL TRIAL: NCT04799002
Title: Choice of Topotecan or Melphalan in Retinoblastoma Patients
Brief Title: Topotecan and Melphalan for Retinoblastoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Huasheng Yang, Principal Investigator, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202103
Record Dates: First submitted 2021-03-12; First posted 2021-03-16 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Retinoblastoma; Chemotherapy Effect
Keywords: Retinoblastoma; topotecan; Melphalan
MeSH Terms: conditions — Retinoblastoma | interventions — Topotecan; Melphalan

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Topotecan (Active Comparator): Topotecan intraocular injection during chemotherapy
  Interventions: Drug: Topotecan
- Melphalan (Experimental): Melphalan intraocular injection during chemotherapy
  Interventions: Drug: Melphalan

INTERVENTIONS:
Drug: Topotecan — Topotecan intraocular injection for chemotherapy in retinoblastoma
  Other Names: Topotecan intraocular injection
  Arms: Topotecan
Drug: Melphalan — Melphalan intraocular injection for chemotherapy in retinoblastoma
  Other Names: Melphalan intraocular injection
  Arms: Melphalan

SUMMARY:
The purpose of this study is to evaluate topotecan and melphalan for retinoblastoma patients.

DETAILED DESCRIPTION:
To evaluate the effectiveness and complications of topotecan and melphalan for intraocular injection in retinoblastoma patients.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed as retinoblastoma
* receiving eyeball-sparing treatment

Exclusion Criteria:

* disease progression during follow-up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-03-11 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Eyeball-sparing rate | 5 years after chemotherapy
  Eyeball-sparing rate during chemotherapy in retinoblastoma patients

SECONDARY OUTCOMES:
Side effects | 5 years after chemotherapy
  Side effects during and after chemotherapy in retinoblastoma patients

CONTACTS AND LOCATIONS:
Overall Officials: Huashen Yang, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No